CLINICAL TRIAL: NCT05204966
Title: Development of Dysphagia Evaluation Via Video Analysis Based on Deep Learning Method in Neonates and Infants and Correlation Between the Evaluation and the Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hong Garam, Director, Principal investigator, Resident of Physical Medicine and Rehabilitation, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S2021-1661-0001
Record Dates: First submitted 2022-01-03; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Dysphagia of Newborn

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infant with suspected dysphagia (Other): For newborns and infants who satisfy the inclusion and exclusion criteria, after taking a video of a bottle feeding, we try to develop an evaluation of swallowing disorder through artificial intelligence-based analysis. The developed evaluation will be verified for validity by comparing it with NOMAS (and VFSS if possible), and the correlation with future development will be analyzed through the relationship with the 1st and 2nd year correctional Bailey Developmental Evaluation.
  Interventions: Diagnostic Test: AI analysis

INTERVENTIONS:
Diagnostic Test: AI analysis — 1. Bottle feeding filming
     - With a camera that can measure depth, take a video of feeding milk from a bottle for 5-10 minutes.
  2. NOMAS (Neonatal Oral-Motor Assessment Scale) evaluation
     * Evaluate NOMAS with bottle feeding video by certified evaluators.
     * NOMAS, developed by Marjorie Meyer Palmer in 1983, is an evaluation method for dysphagia applicable to infants under 48 weeks of PMA.
  3. Implementation of video analysis using deep learning (A) Analysis method - Implement a deep learning network that sets keypoints of faces and environments related to swallowing and detects specified keypoints in units of frames.
  (B) Analyze the movement of key points, and figure out the correlation between swallowing states.
  (C) Create an input/output process that can automatically classify swallowing states with video as input.

SUMMARY:
The purpose of this study is to develop an evaluation of dysphagia through deep learning-based video analysis in newborns and infants, and to report the correlation with future development.

DETAILED DESCRIPTION:
Although the exact frequency of dysphagia in newborns is not known, according to a paper published by Motion et al. in 2001, the prevalence of eating problems in premature infants under 37 weeks of age was 10.5%, and in 2001, Mercado-Deane et al. reported that about 26% had dysphagia. In 1996, Reilly et al. reported that more than 90% of children with polio had oral movement disorders and 38% had dysphagia. It is known that the frequency of dysphagia in newborns and infants is not low. The risk factors that cause these dysphagia are very diverse, and dysphagia in children can be induced by causes that can affect the whole process of swallowing.

The evaluation of dysphagia can be divided into an evaluation method that does not use an instrument such as SOMA, SDS, and quality of life measurement, and an evaluation method that uses an instrument such as VFSS and FEES. However, it is difficult to conduct tests such as VFSS in newborns and infants due to poor coordination, and there is also a risk of radiation exposure. In addition, there are practical difficulties in applying the evaluation in all medical institutions because special facilities are required to implement VFSS and specialized clinical personnel are required.

The Neonatal Oral-Motor Assessment Scale (NOMAS), developed by Marjorie Meyer Palmer in 1983, is an evaluation method for dysphagia applicable to infants under 48 weeks of PMA that evaluates whether there are abnormal findings by observing sucking for 5 minutes. However, NOMAS has the disadvantage that a person has to directly observe the sucking and may show differences in results between raters.

Therefore, in this study, inspired by the evaluation method of NOMAS, investigators try to develop an evaluation method to evaluate swallowing disorders by videotaping bottle feeding in newborns and infants, then calculating and analyzing the features of the baby's face related to swallowing with artificial intelligence. investigators would like to analyze the relationship between this evaluation result and future development.

ELIGIBILITY:
Inclusion Criteria:

* Newborns and infants under 6 months of correctional age
* Clinically suspected to have dysphagia
* In case parental consent is obtained

Exclusion Criteria:

* In case of cardiopulmonary instability (ECMO, Ventilator, etc. are being applied)
* When it is not possible to secure sufficient fields for artificial intelligence analysis of images due to factors such as anatomical abnormalities of the head and neck

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between NOMAS evaluation and AI analysis of dysphagia | up to 2 years
  Correlation between NOMAS evaluation and AI analysis of dysphagia
Correlation between VFSS evaluation and AI analysis of dysphagia | up to 2 years
  Correlation between VFSS evaluation and AI analysis of dysphagia

SECONDARY OUTCOMES:
Correlation between AI analysis of dysphagia and development | up to 2 years
  Correlation between AI analysis of dysphagia and development

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided